CLINICAL TRIAL: NCT05840939
Title: The Effect of Pranayama and Diaphragmatic Breathing Exercise on Sleep Quality, Pain and Fatigue Level in Female Patients With Fibromyalgia
Brief Title: Pranayama and Diaphragmatic Breathing Exercise Applied to Female Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Meltem Sungur, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2344633
Record Dates: First submitted 2023-04-06; First posted 2023-05-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Pranayama; Diaphragmatic breathing; Quality of sleep; Pain; Fatigue
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders; Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: This study was conducted as a single-blind randomized controlled study with pretest-posttest.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pranayama (Experimental): At the beginning, each patient in this group was shown one-on-one by the researcher and taught by applying them together, taking into account the application steps, how to practice pranayama. In the next step, the patients were asked to do this application themselves. Sleep quality, pain and fatigue levels of the patients were determined after 6 weeks.
  Interventions: Behavioral: Pranayama
- diaphragm breathing exercise group (Experimental): At the beginning, the patients in this group were shown how to do the diaphragm breathing exercise and how to do the diaphragm breathing exercise, taking into account the application steps, each patient was shown individually by the researcher and taught by applying them together. In the next step, the patients were asked to do this application themselves. Sleep quality, pain and fatigue levels of the patients were determined after 6 weeks.
  Interventions: Behavioral: diaphragm breathing exercise
- control group (No Intervention): It is the group where no application has been made.

INTERVENTIONS:
Behavioral: Pranayama — Pranayama, one of the practices of yoga, is a Sanskrit word consisting of a combination of two words, a technique of rhythmic, controlled breathing. So "prana" means life breath/life energy and "ayama" means expansion/regulation/control. Pranayama helps to improve lung capacity, heart and respiratory functions, nervous and hormonal systems, as well as mental activity.
  Arms: pranayama
Behavioral: diaphragm breathing exercise — Diaphragmatic breathing is also known as deep breathing or slow abdominal breathing. This breathing exercise uses the diaphragm muscle. The diaphragm is the muscle under the lungs that supports the lungs in up and down breathing.
  Arms: diaphragm breathing exercise group

SUMMARY:
Female patients diagnosed with fibromyalgia were divided into pranayama breathing exercise, diaphragm breathing exercise and control groups. The sleep quality, pain and fatigue levels of the patients in the intervention group were determined before and after the breathing exercise.

DETAILED DESCRIPTION:
Aim: This study was conducted to determine the effect of pranayama and diaphragm breathing exercises applied to female patients diagnosed with fibromyalgia on sleep quality, pain and fatigue levels.

Material and Method: This study, designed as a randomized controlled and experimental study, was conducted between November 2022 and June 2023. The data of the study consisted of 100 female patients diagnosed with fibromyalgia: 32 in the pranayama group, 33 in the diaphragm breathing exercise group and 35 in the control group. As data collection tools; Patient Information Form, Visual Analog Scale, Fatigue Severity Scale and Pittsburgh Sleep Quality Scale were used. During the study, the control group received routine treatment, while the two groups in the intervention group received the following training given by the researcher; They were asked to do pranayama and diaphragm breathing exercise 3 sets a day (morning-afternoon-evening), 7 days a week for 6 weeks. At the end of this process, sleep quality, pain and fatigue levels of three groups were evaluated again.

Results: It was observed that there was no statistically significant difference between the initial pain and sleep quality total scores of three groups (p>0.05), there was a significant difference between the groups in terms of pain, fatigue and sleep quality scores after the application (p<0.05).

Conclusion: As a result, it was determined that breathing exercises reduced the patients' pain and fatigue levels and improved their sleep quality.

Keywords: Pain, diaphragmatic breathing, fibromyalgia, pranayama, sleep quality, fatigue

ELIGIBILITY:
Inclusion Criteria:

•● Being 18 years or older

* Being a female patient who has had pain for at least three months and has been diagnosed with fibromyalgia by a physician according to the ACR 2016 fibromyalgia diagnostic criteria.
* Having a PSQI score of five and above
* Complaint of fatigue and getting a score of 4 or above on the fatigue severity scale
* Pain score of one or above according to VAS
* Having no communication problems and knowing how to read, write and speak Turkish
* Not being pregnant and not breastfeeding

Exclusion Criteria:

* Having a malignancy related to the respiratory system (bronchus or lung)
* Having tuberculosis disease
* Having chest pain
* Having any psychiatric diagnosis during outpatient clinic screenings
* Having a nasal septum derivation or adenoid that will affect the ventilation process
* Having previously practiced/trained in pranayama or diaphragmatic breathing exercises

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being female
Enrollment: 100 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | [Time Frame: 6 weeks]
  "0" indicates no pain and "10" indicates the most severe level of pain. On the scale, <3 mild pain, 3-6 moderate pain, >6 severe pain were specified.

CONTACTS AND LOCATIONS:
Overall Officials: MELTEM SUNGUR, Principal Investigator — Kilis 7 Aralik University
Locations (1):
- Meltem Sungur, Şahinbey, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Can be reviewed by other researchers after the study has been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: data will be shared as long as they are published
Access Criteria: publication page